CLINICAL TRIAL: NCT04680182
Title: Axillary and Inguinal Lymph Node Dissection in Stage III Melanoma Patients: A Prospective Randomized Trial of Two Approaches to Wound Drainage
Brief Title: Early Complications After Axillary and Inguinal Lymph Node Dissection in Stage III Melanoma Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Lars Frich, Consultant in general and plastic surgery, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-07777
Record Dates: First submitted 2020-12-17; First posted 2020-12-22 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-09

CONDITIONS: Melanoma; Complication
Keywords: Melanoma; Complication; Drain; Non-inferior study; Randomized study; Seroma
MeSH Terms: conditions — Melanoma; Seroma

STUDY DESIGN:
Intervention Model Description: Non-inferiority randomised study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Wound drain is kept until until a scheduled visit three weeks after the surgery unless the drain produced less than 30 ml/day for two consecutive days, in which case it could be removed earlier.
  Interventions: Procedure: Suction drain
- Control group (Active Comparator): When the drain produces less than 100 mL over 24 hours, the self-suction bulb is removed and the drain is shortened and drained into a colostomy bag placed around the site of drain insertion. A request is filed with the community nursing system to have a visiting nurse to pull out the drain 1-2 cm per day.
  Interventions: Procedure: Suction drain

INTERVENTIONS:
Procedure: Suction drain — Suction drain either kept for three weeks or gradually pulled out.

SUMMARY:
This prospective randomized non-inferiority study is designed to compare the rate and severity of complications after axillary and inguinal lymph node dissection in stage III melanoma patients in a study group where the drain is left in place for three weeks and a control group consisting of patients managed according to the standard institutional protocol. Furthermore, variables associated with complications will be examined.

DETAILED DESCRIPTION:
Consecutive stage III melanoma patients 18 years or older referred to our institution for axillary or inguinal lymph node dissection is eligible for inclusion of the study. A bipolar vessel sealing device (LigaSure, Covidien) will be used for dissection in all procedures. All patients will be scheduled for an outpatient visit with an experienced nurse three weeks after the surgery. Any deviation from the normal postoperative course will be recorded in the electronic patient journal. Complications are graded according to the Clavien-Dindo classification. Patients with complications or with suspected complications at the three-week follow up will be scheduled for new an outpatient visit. Patient demographics, clinicopathological characteristics of the primary melanoma, indication for the procedure, length of postoperative stay and early complications and treatment for complications will be collected for analysis

ELIGIBILITY:
Inclusion Criteria:

* stage III melanoma patients with confirmed metastases to lymph nodes in axilla or groin

Exclusion Criteria:

* unable to follow instructions or provide an informed written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2018-05-11 (Actual); Primary Completion 2021-04-06 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Non-inferiority of overall early complications | 3-week follow up, total 3 months
  To determine if the study group was non-inferior to the control group

SECONDARY OUTCOMES:
Rate and severity of early complications | 3-week follow up, total 3 months
  Frequency of each complication and an analysis of possible risk factors.

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Oslo, Norway